CLINICAL TRIAL: NCT02114567
Title: Neural Triggering and Cycling-off of Pressure Support Ventilation Improves Synchrony and Reduces Inspiratory Effort in Chronic Obstructive Pulmonary Disease.
Brief Title: Is it Necessary to Set External PEEP in AECOPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Dr., Southeast University, China
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: COPDNAVA
Record Dates: First submitted 2013-11-04; First posted 2014-04-15 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Acute Exacerbation Chronic Obstructive Pulmonary Disease
Keywords: AECOPD; work of breathing; patient-ventilator synchrony

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PSV ventilation (Experimental): AECOPD Patients who were ventilated wiht PSV, PEEP was titrated and set at 0, 40%, 80% and 120% PEEPi. Pressure support was set to get the tidal volume of 6ml/kg.
  Interventions: Other: PEEP titration
- NAVA ventilation (Experimental): AECOPD patients who were ventilated with NAVA, PEEP was titrated and set at 0, 40%, 80% and 120% PEEPi. NAVA level was set to get the tidal volume of 6ml/kg.
  Interventions: Other: PEEP titration

INTERVENTIONS:
Other: PEEP titration — In both groups, PEEP was titrated and set to 0, 40%PEEPi, 80%PEEPi, and 120%PEEPi

SUMMARY:
Acute exacerbation of chronic obstructive pulmonary disease patients with intrinsic positive end-expiratory pressure (PEEPi), Neurally adjusted ventilatory assist (NAVA) reduce work of breathing and trigger delay at any external positive end-expiratory pressure (PEEPe) level compared with pressure-support ventilation (PSV)

DETAILED DESCRIPTION:
All patients randomly underwent a 30 mins PSV and NAVA crossover ventilation (15 mins each) at progressive PEEPe levels. Progressive levels of PEEPe were applied stepwise in increments of 40% of baseline static PEEPi, every 30 mins, from zero to 160% of baseline static PEEPi during the protocol (0, 40%, 80%, 120% and 160% of static PEEPi, respectively). During PSV, pressure support level was set to meet a Vt 6ml/kg, I/E cycling was 30% of the maximum inspiratory peak flow, flow trigger was 1L/min, and inspired fraction of oxygen (FiO2) was set to the similar level before the study protocol. During NAVA, NAVA Level was set at 15 cmH2O / µV and a peak airway pressure limit was set in order to apply the same inspiratory pressure support at each PEEPe level during PSV. The new setting of NAVA was defined as NAVA15. Moreover the trigger was set at 0.5 µV and the I/E cycling fixed at 70% of the peak of EAdi. During the entire protocol, FiO2 and peak air way pressure were maintained the same levels at each PEEPe level between PSV and NAVA. Arterial blood gases were measured at the end of PSV or NAVA15 ventilation at each PEEPe level.

ELIGIBILITY:
Inclusion Criteria:

1. mechanical ventilation AECOPD patients with Static PEEPi measured by End-expiratory airway occlusion method ≥ of 5 cm H2O
2. Hemodynamics stability (heart rate < 140 beats/min, no vasopressors required, or <5 μg/kg/min dopamine) without any evidence
3. no sedation or on minimal sedation with low dose of morphine (<3mg/h, by continuous intravenous infusion
4. Breathing spontaneously
5. Awake and with positive cooperate

Exclusion Criteria:

1. tracheostomy
2. treatment abandonment
3. history of esophageal varices
4. gastro-esophageal surgery in the previous 12 months or gastro-esophageal bleeding in the previous 30 days
5. coagulation disorders (INR ratio>1.5 and Activated partial thromboplastin time > 44 s)
6. history of acute central or peripheral nervous system disorder or severe neuromuscular disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
trigger work of breathing | 1 day

SECONDARY OUTCOMES:
patient-ventilator synchrony | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: ling liu, md, Study Director — Department of Critical Care Medicine, Nanjing Zhongda Hospital and School of Medicine, Southeast University, China
Locations (1):
- Nanjing Zhong-Da Hospital, Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Liu L, Xia F, Yang Y, Longhini F, Navalesi P, Beck J, Sinderby C, Qiu H. Neural versus pneumatic control of pressure support in patients with chronic obstructive pulmonary diseases at different levels of positive end expiratory pressure: a physiological study. Crit Care. 2015 Jun 9;19(1):244. doi: 10.1186/s13054-015-0971-0. PMID 26059238